CLINICAL TRIAL: NCT00606918
Title: Validation of a New Device to Measure Neuromuscular Disease Progression
Acronym: ATLIS
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Patricia L. Andres, Massachusetts General Hospital
Other Study IDs: MDA-4343
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Amyotrophic Lateral Sclerosis & Other Neuromuscular Disorders
Keywords: Strength testing; Disease progression; ALS; Healthy Adults
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Individuals with ALS
- 2: Healthy Adults

SUMMARY:
There is a great need for the development of sensitive outcomes that allow experimental drugs to be tested in human subjects more efficiently. If we could more precisely measure whether an experimental drug slows the progression of ALS or other neuromuscular diseases, this would allow more drugs to be tested quicker and at less expense. We have developed a new device that accurately measures isometric strength called: Accurate Test of Limb Isometric Strength (ATLIS). This device was designed to be portable, quick, and easy to use, while generating accurate and reliable, interval level data. This study will enable us to test the reliability and validity of ATLIS.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be at least 18 years old and able to provide informed consent
* All subjects have no health conditions that limit their ability to safely exert maximal force using the muscles in their arms and legs.
* Subjects with a diagnosis of laboratory supported probable, probable or definite ALS according to the World Federation of Neurology El Escorial, as determined by their referring neurologist at MGH.
* All subjects must be able to speak and understand English.

Exclusion Criteria:

* Presence of significant arthritis, orthopedic conditions, or cardio-pulmonary conditions or other medical conditions that may limit the ability to maximally exert force safely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with ALS
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
isometric strength measures | cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L. Andres, MS, DPT, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - East, Charlestown, Massachusetts, United States